CLINICAL TRIAL: NCT04788160
Title: Effects of Cervical SNAG Half Rotation Technique in Cervicogenic Headache Patients.
Brief Title: Cervical SNAG Half Rotation Technique in Cervicogenic Headache Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00765 Yusra javed
Record Dates: First submitted 2021-02-16; First posted 2021-03-09 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Cervicogenic Headache
Keywords: SNAGs; cervicogenic headache; FRT; NDI; NPRS
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical SNAGs along with conventional therapy (Experimental): patient will receive Cervical SNAGs along with conventional therapy (Group A)
  Interventions: Other: Cervical SNAGs along with conventional therapy
- Conventional Therapy (Other): patient will receive only conventional therapy (Group B)
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Cervical SNAGs along with conventional therapy — cervical SNAG half rotation technique will be performed with the patient sitting on a chair in the erect posture. The therapist placed his thumb over thumb over the transverse process of C1. Then, he glided ventrally with active rotation of the restricted site 10 times holding for 10 seconds with overpressure at end of the rotation with 30 second rest in between each repetition and 3 session/week for 4 weeks.
  * Conventional therapy will include:
  * Hot pack over the cervical region for 10 minutes.
  * TENS for 10 minutes.
  * Furthermore, general stretching the upper cervical muscles will be done with 5 repetitions with 3 sessions/week for 4 weeks.
  * Isometric cervical extensor exercise with 10 seconds hold for 10 times will be done.
  * Cervical flexor strengthening will be done 10 times in sitting position.
  Arms: Cervical SNAGs along with conventional therapy
Other: Conventional Therapy — * Patients in this group will undergo only conventional therapy which will include:
  * Hot pack for 15 minutes.
  * TENS for 10 minutes.
  * Furthermore, general stretching the upper cervical muscles will be done with 5 repetitions each 3 sessions/week for 4 weeks.
  * Isometric cervical extensor exercise with 10 seconds hold for 10 times will be done.
  * Cervical flexor strengthening will be given to the patient by the therapist, 10 times in sitting position.
  Arms: Conventional Therapy

SUMMARY:
The purpose of this study is to find out the effect of cervical sustained natural apophyseal glide half rotation technique in patients with cervicogenic headache. Not many researches have focused specifically on the cervical sustained natural apophyseal glide half rotation technique and this study intends to see its effect in the cervicogenic headache patients.

DETAILED DESCRIPTION:
Cervicogenic headache is a very frequent complaint that is commonly faced by general population. The International Headache Society placed cervicogenic headache in the secondary headache sub-group. The global prevalence of headache is about 47%, whereas 15% to 20% of those are Cervicogenic headache .Females are four times more prone to Cervicogenic headache than males. Persons with chronic Cervicogenic headache experience significant restriction of everyday function and are limited to social involvement, and emotional sufferings. Beside this, the poorer quality of life is seen in these individuals than normal. Headache can be classified as primary or secondary. Primary headache originates from a vascular or muscular source such as tension-type headache. Secondary headache is related to other structures with cervicogenic headache being the most common type that is related to cervical spine dysfunction. Up to about 70% of frequent intermittent headache are reported with associated neck pain making cervicogenic headache difficult to diagnose.

The C1-C2 segment is considered essential to be examined in Cervicogenic headache diagnosis. Moreover, muscle tightness especially of the upper trapezius and sternocleidomastoid muscles with impaired strength and neuromotor contract of the cervical flexors (superficial and deep) are frequently encountered in subjects with Cervicogenic headache. Different therapeutic approaches have been proposed for treatment of headaches; with physical therapy, pharmacological drugs, and cognitive therapies most commonly used. Several studies reported that manual therapy of the cervical spine can decrease pain intensity, frequency, and duration in addition to reduction in neck pain and disability. The "mobilization with movement" concept, known as the Mulligan concept, is entirely distinct from other forms of manual therapy. Mulligan described the sustained natural apophyseal glide on the joint with active movement done by the patient in the direction of the symptoms. This glide should be pain-free, with proper force applied by a trained person.

The efficacy of sustained natural apophyseal glide C1-C2 has been proven in a research in patients who were experiencing acute to subacute Cervicogenic headache for both short and long-term periods. Mulligan recommended that mobilization should be done towards the restricted site or in the direction of symptom reproduction, which is difficult to find in patients experiencing headache and dizziness in only one direction. There is evidence that mobilizing symptomatic and asymptomatic cervical levels results in immediate improvement of pain and segmental mobility at the same level as well as adjacent areas. sustained natural apophyseal glide Mulligan mobilizations are one of the most popular manual therapy techniques found to be effective in treating Cervicogenic headache as mentioned in the "Neck Pain Guidelines 2017" recommended by American Physical Therapy Association , which reported that patients with neck pain and Cervicogenic headache had significant improvement with self-sustained natural apophyseal glide C1-C2 for both short and long-term periods.

Additionally, sustained natural apophyseal glide as a treatment modality can be applied to all the spinal joints, the rib cage and the sacroiliac joint. They provide a method to improve restricted joint range when symptoms are movement induced. The therapist facilitates the appropriate accessory zygoapophyseal joint glide while the patient performs the symptomatic movement. The facilitatory glide must result in full-range pain-free movement. Sustained end range holds or overpressure can be applied to the physiological movement. This previously symptomatic motion is repeated up to three times while the therapist continues to maintain the appropriate accessory glide. In particular, a cervical sustained natural apophyseal glide is applied with the patient seated, and thus, the spine is in a vertical (i.e. weight bearing or loaded) position.

Mobilization is very effective in the management of Cervicogenic headache. The group of patients who are given sustained natural apophyseal glide showed significantly greater improvement in neck disability index. A research study has shown that the headache sustained natural apophyseal glide is more effective as compared to the reverse headache sustained natural apophyseal glide in the reduction of pain on headache scale. Another research study has shown that C2 sustained natural apophyseal glide and reverse sustained natural apophyseal glide technique were effective in reducing functional disability and headache intensity. Also, C2 sustained natural apophyseal glide was found to be more effective in reducing headache intensity when compared with the other group.

ELIGIBILITY:
Inclusion Criteria:

* Patients having experienced headache in the last three months and those with unilateral neck pain.
* Patients experiencing stiffness are also included along with those exhibiting limited range of motion of neck >10 degree which will be confirmed positive through FRT (flexion-rotation test).

Exclusion Criteria:

* Congenital conditions of the cervical spine
* Disc herniation patients or fractures in the cervical spine.
* VBI and associated dizziness
* Vestibular dysfunctions.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 12th day
  This scale will be used for assessing low back pain before and after treatment.0 no pain 1-4 mild pain 5-7 moderate and 8-10 sever pain. Baseline,6th day and 12th day
Flexion rotation test (FRT) | 12th day
  The cervical flexion-rotation test (FRT) is used to assist in the diagnosis of CGH and, in particular, C1-C2 segmental dysfunction.Normal range of movement is 44° to each side. The reliability of the test is ICC= 0.7 to 0.75 along with 95% confidence interval
Neck disability index (NDI) | 12th day
  gives information about how much neck pain affects the ability to manage everyday life. The reliability of this test in Urdu version is ICC= 0.50 to 0.98

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Umar M, Naeem A, Badshah M, Zaidi S. A randomized control trial to review the effectiveness of cervical mobilization combined with stretching exercises in cervicogenic headache. J Public Health Biolo Sci. 2012;1(1):09-13.
- [Background] Hall T, Briffa K, Hopper D. Clinical evaluation of cervicogenic headache: a clinical perspective. J Man Manip Ther. 2008;16(2):73-80. doi: 10.1179/106698108790818422. PMID 19119390
- [Background] Petersen SM. Articular and muscular impairments in cervicogenic headache: a case report. J Orthop Sports Phys Ther. 2003 Jan;33(1):21-30; discussion 30-2. doi: 10.2519/jospt.2003.33.1.21. PMID 12570283
- [Background] Islam R, Quddus N, Miraj M, Anwer S. Efficacy of deep cervical flexor strength training versus conventional treatment in cervicogenic headache. Int J Cur Res Rev. 2013;5(08):84-90.
- [Background] Fernandez-de-Las-Penas C, Courtney CA. Clinical reasoning for manual therapy management of tension type and cervicogenic headache. J Man Manip Ther. 2014 Feb;22(1):44-50. doi: 10.1179/2042618613Y.0000000050. PMID 24976747
- [Background] Garcia JD, Arnold S, Tetley K, Voight K, Frank RA. Mobilization and Manipulation of the Cervical Spine in Patients with Cervicogenic Headache: Any Scientific Evidence? Front Neurol. 2016 Mar 21;7:40. doi: 10.3389/fneur.2016.00040. eCollection 2016. PMID 27047446
- [Background] Teys P, Bisset L, Vicenzino B. The initial effects of a Mulligan's mobilization with movement technique on range of movement and pressure pain threshold in pain-limited shoulders. Man Ther. 2008 Feb;13(1):37-42. doi: 10.1016/j.math.2006.07.011. Epub 2006 Oct 27. PMID 17070090
- [Background] Gross A, Kay TM, Paquin JP, Blanchette S, Lalonde P, Christie T, Dupont G, Graham N, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Hoving JL, Bronfort G, Santaguida PL; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2015 Jan 28;1(1):CD004250. doi: 10.1002/14651858.CD004250.pub5. PMID 25629215
- [Background] Slaven EJ, Goode AP, Coronado RA, Poole C, Hegedus EJ. The relative effectiveness of segment specific level and non-specific level spinal joint mobilization on pain and range of motion: results of a systematic review and meta-analysis. J Man Manip Ther. 2013 Feb;21(1):7-17. doi: 10.1179/2042618612Y.0000000016. PMID 24421608
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Wilson E. The Mulligan concept: NAGS, SNAGS and mobilizations with movement. Journal of Bodywork and Movement Therapies. 2001;5(2):81-9.
- [Background] Exelby L. The Mulligan concept: its application in the management of spinal conditions. Man Ther. 2002 May;7(2):64-70. doi: 10.1054/math.2001.0435. PMID 12374089